CLINICAL TRIAL: NCT00195429
Title: A Randomized, Open-label and Multicenter Trial Comparing Withdrawal of Steroids or Tacrolimus From Sirolimus-based Immunosuppressive Regimen in de Novo Renal Allograft Recipients
Brief Title: A Study Comparing the Withdrawal of Steroids or Tacrolimus in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E-101535
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2010-04

CONDITIONS: Kidney Failure; Graft vs Host Disease
Keywords: Kidney; Transplant
MeSH Terms: conditions — Renal Insufficiency; Graft vs Host Disease | interventions — Tacrolimus; Sirolimus; Prednisone

ARMS (2):
- Sirolimus + Tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus; Drug: Sirolimus
- Sirolimus + Prednisone (Active Comparator)
  Interventions: Drug: Sirolimus; Drug: prednisone

INTERVENTIONS:
Drug: Tacrolimus
  Arms: Sirolimus + Tacrolimus
Drug: Sirolimus
Drug: prednisone
  Arms: Sirolimus + Prednisone

SUMMARY:
This study evaluates two different immunosuppression drug regimens in patients with a recent kidney transplant. Patients initially received a regimen of Sirolimus, Tacrolimus and Prednisone and then randomized to discontinue either Tacrolimus or Prednisone.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease, with patients scheduled to receive a kidney transplant.
* Women who are of childbearing potential who are not pregnant and agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation of study drugs. Any woman becoming pregnant during the treatment period must discontinue the use of study drugs;
* Signed informed consent.

Exclusion Criteria:

* Evidence of active systemic or localized major infection at the time of initial study drug administration;
* Multiple organ transplants;
* Any pathology or medical condition that can interfere with this protocol study proposal.

Other exclusion applies.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-08; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com
Locations (1):
- São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Brazil from August 2005 to September 2006.
Pre-assignment Details: After renal transplantation subjects were immediately randomized into day 1.
Period: Overall Study
Arm/Group | Sirolimus + Tacrolimus | Sirolimus + Prednisone
Started | 24 | 23
Completed | 19 | 18
Not Completed | 5 | 5
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus + Tacrolimus | Sirolimus + Prednisone | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.3) | 34.7 (12.2) | 35.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Biopsy Confirmed Acute Rejection at 12 Months Follow up.
Description: Diagnosis of acute rejection was made via kidney biopsy using the Banff criteria (a standardized model for interpretation of renal allograft biopsies).
Time Frame: 12 months
Population: The population that was used for this analysis was the transplantation recipient population, which included all randomized patients.
Measure: Number; unit: participants
Arm/Group | Sirolimus + Tacrolimus | Sirolimus + Prednisone
Number analyzed (Participants) | 24 | 23
participants
  Subjects with Acute Rejection | 3 | 3
  Subjects without Acute Rejection | 21 | 20
Statistical Analysis 1: Comparison: Sirolimus + Tacrolimus vs Sirolimus + Prednisone; Test type: Superiority or Other; p = 1.0, Fisher Exact

2. Secondary Outcome: Creatinine Clearance Rate
Description: Creatinine clearance is a measure of kidney function. Creatinine clearance rate (CCr) is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Creatinine clearance can be measured directly or estimated using established formulas. For this study, CCr was calculated using the Nakivell formula. Normal values for healthy, young males are in the range of 100-135 ml/min and for females, 90-125 ml/min. Creatinine clearance decreases with age. A low creatinine clearance rate indicates poor kidney function.
Time Frame: 12 months
Population: The population that was used for this analysis was patients who completed 12 months.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Sirolimus + Tacrolimus | Sirolimus + Prednisone
Number analyzed (Participants) | 19 | 18
ml/min | 60 (11.5) | 63.4 (10.5)
Statistical Analysis 1: Comparison: Sirolimus + Tacrolimus vs Sirolimus + Prednisone; Test type: Superiority or Other; p = 0.361, Student's t-test

ADVERSE EVENTS:
Arm/Group | Sirolimus + Tacrolimus | Sirolimus + Prednisone
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 23/24 | 22/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus + Tacrolimus (N=24) | Sirolimus + Prednisone (N=23)
Infection Disease (Infections and infestations) | 19 | 19
Hypertension (Vascular disorders) | 1 | 1
Diabetes Mellitus post-transplant (Metabolism and nutrition disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.